CLINICAL TRIAL: NCT07074262
Title: Comparison Between the Effect of Dexmedetomidine _midazolam and ketamine_midazolam Combination on Post Operative Delirium and Cognitive Disorders in Cardiac Patients Undergoing non_cardiac Surgery
Brief Title: Comparison Between the Effect of Dexmedetomidine _midazolam and ketamine_midazolam Combination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hanaa Fathy Mohamed, Specialist of Anesthesia, intensive care and pain management,Faculty of Medicine, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hanaa Fathy Mohamed
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Cognitive Dysfunction; Post Operative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): About 38 participants received conventional general anesthesia only. Smooth Induction of anesthesia will be done by injecting fentanyl 3-5 μg/kg IV - Midazolam 0.05 to 0.15 mg/kg(Dormicum 1mg/1m ampoul AMOUN com) to be titrated (and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine gel 2 %. Maintenance of anesthesia will be done using sevoflurane 1.5-2 %, and Mixture of O2 and Air (70%:30%).
  Interventions: Drug: Ketamine
- Ketamine group (Active Comparator): About 38 participants received conventional general anesthesia with administration of Ketamine before induction as follow: Ketamine 1 mg /kg(ketalar Vial 50mg/ml pfzer com) will be administered IV before induction, then a smooth Induction of anesthesia will be done by injecting fentanyl 3-5 μg/kg(23) Midazolam 0.05 to 0.15 mg/kg to be titrated (24) and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine gel 2 %. Maintenance of anesthesia will be done using sevoflurane 1.5-2% and mixture of O2 and Air (70%: 30%).
  Interventions: Drug: Ketamine
- Dexmedetomidine group (Active Comparator): About 38 participants received conventional general anesthesia with administration of dexmedetomidine before induction as follow:Dexmedetomidine(precedex 100mc/ml 1 mcg Pfizer com) will be injected IV before Induction of anesthesia. Then Induction of anesthesia will be done by injecting fentanyl 3-5 μg/kg(23), Midazolam 0.05 to 0.15 mg/kg to be titrated (24) and atracurium 0.5 mg/kg for muscle relaxation. Laryngoscopy and endotracheal intubation will be performed using oral cuffed tube lubricated with lidocaine gel 2 %. Maintenance of anesthesia will be done using sevoflurane 1.5-2% and mixture of O2 and Air (70%: 30%).
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — to compare the effect of Ketamine versus Dexmedetomidine on postoperative cognitive dysfunction and delirium in all cardiac patient undergoing low risk non-cardic surgery.
  Other Names: Dexmedetomidine

SUMMARY:
Postoperative cognitive dysfunction (POCD) is one of the most common complications after anesthesia, with a prevalence of approximately 12% and a higher prevalence of up to 41.4% in older surgical patients during the entire hospitalization period .A variety of pharmacological therapies are utilized to prevent or minimize POCD.

Post-operative delirium is also one of the most common complications following anaesthesia with frequency estimates ranging from 10 to 50%. It is defined as delirium occurring 24 to 72 hours after surgery. There are multiple risk factors for developing postoperative delirium including pre-existing dementia, old age, medical co-morbidities, and psycopathological symptoms.

The recognition and treatment of Post-operative delirium is critically important because postoperative delirium is associated with poor outcomes including functional decline, dementia, cognitive impairment, increased hospital length of stay , increased mortality ( 11% increasing in the risk of death at 3 months and up to a 17% increased risk of death at 1 year. Previous studies have examined the relationship between patient-related factors, surgical factors and postoperative delirium.

Few studies have examined events in the postoperative period that may contribute to the occurrence of postoperative delirium. Two related and possibly modifiable factors in the postoperative period are postoperative pain and analgesic medications. Although prior studies suggest that postoperative pain and analgesia are associated with postoperative delirium.

DETAILED DESCRIPTION:
POCD) is a subtle disorder of thought processes, which may influence isolated domains of cognition such as verbal memory, visual memory, language comprehension, visuospatial abstraction, attention, or concentration.It is to be distinguished from postoperative delirium, which tends to be a transient and fluctuating disturbance of consciousness that tends to occur shortly after surgery, whereas POCD is a more persistent problem of a change in cognitive performance as assessed by neuropsychological tests.

Delirium is defined by the Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV) as an acute and fluctuating disturbance in consciousness that may or may not be accompanied by agitation.Delirium has been reported to occur in 10% to 60% of surgical patients, however, the incidence of delirium in older surgical patients may be as high as 73% depending on the diagnostic method used.

Acute post-surgical pain leads to delayed discharge from post-operative recovery area, impairs pulmonary and immune functions, increases risk of ileus, thromboembolism, myocardial infarction and may lead to increased length of hospital stay. It is also an important factor leading to the development of chronic persistent post-operative pain in almost half of the patients.

Acute postoperative pain remains one of the major challenges of pain medicine. Although various methods and drugs have been proposed to manage perioperative pain, oral and intravenous opioid analgesics are still among the most common medications. However, their potential short-and long-term adverse effects can limit their application.

Dexmedetomidine is an alpha-2 adrenoceptor agonist with analgesic and neuroprotec-tive effects. These neuroprotective characteristics may explain the growing evidence of the preventative effect of dexmedetomidine on POCD.

Ketamine, which is a dissociative anaesthetic, is having all the properties which we needed i.e. an intravenous anesthetic with distinct analgesic activity and relatively rapid onset of action with immediate recovery. The precise molecular mechanism of ketamine has been extensively studied during the last decade and the current understanding is that inhibition of sensory perception is mediated by the blockade of N-methyl D-aspartate receptor blockade.

ELIGIBILITY:
Inclusion Criteria:

* ASA (II - III) patients above 40 years old.
* Patients diagnosed with a cardiac condition (coronary artery disease, Valvular heart disease , arrhythmias, hypertension ) with EF > 40% and Moderate to good functional capacity (METS > 4).
* Patients scheduled to undergo low risk non-cardiac surgical procedures

Exclusion Criteria:

* Patients having gross hemodynamic or ventilatory fluctuations during the operation.
* Patients with recent myocardial infarction
* Patients who develop postoperative shock, major bleeding or complications.
* Patients with a history of psychiatric disorders.
* Patients with a current history of illicit drug use.
* Patients using hypnotic, anxiolytic, or antipsychotic drugs.
* Allergy to any of the drugs that were used in the study.
* Emergency surgery of Moderate to high risk surgery.
* Pregnancy.
* Patient refusal to give consent

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Cognitive Dysfunction and Delirium | First 24 hours and 48 hours after surgery
  Assessment of the patients whom subjected surgery by using Memorial delirium assessment scale (MDAS) as follows: 1, awareness; 2, orientation; 3, short-term memory; 4, digit span; 5, attention capacity; 6, organizational thinking; 7, perceptual disturbance; 8, delusions; 9, psychomotor activity; and 10, sleep-wake cycle

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Attia Nassef, Professor, Study Chair — Anaesthesiology,Surgical intensive care and pain management,Faculty of Medicine,Beni-Suef University
Locations (1):
- Beni- Suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided